CLINICAL TRIAL: NCT07000097
Title: Use of Three-Dimensional Printed Models for Endovascular Planning and Follow-up in Patients Affected by Aorto-Iliac-Femoral-Popliteal Arterial Disease Undergoing Balloon Angioplasty: Applicability, Effectiveness in Technical Success and on Mid-Term Outcomes, Cost-Analysis, and Exploration of New Technologies. A Single-center, Single-blind Randomized Controlled Trial
Brief Title: Use of Three-Dimensional Printed Models for Endovascular Planning and Follow-up in Patients Affected by Aorto-Iliac-Femoral-Popliteal Arterial Disease Undergoing Balloon Angioplasty. A Single-center, Single-blind Randomized Controlled Trial
Acronym: 3DPAD-1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Paolo Perini, Professor, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR-2019-12369941
Record Dates: First submitted 2025-05-23; First posted 2025-06-02 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Artery Disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative planning performed based on CTA (standard of care) (Active Comparator)
  Interventions: Device: PTA (Standard of Care)
- Preoperative planning performed using CTA and a patient-specific, custom-made 3D-printed model (Experimental)
  Interventions: Device: PTA planning supported by 3D-printed model

INTERVENTIONS:
Device: PTA planning supported by 3D-printed model — Custom-made 3D-printed model as an additional tool to computed tomography angiography for planning Percutaneous Transluminal Angioplasty in aorto-iliac-femoral-popliteal artery disease
  Arms: Preoperative planning performed using CTA and a patient-specific, custom-made 3D-printed model
Device: PTA (Standard of Care) — Preoperative planning performed based on computed tomography angiography
  Arms: Preoperative planning performed based on CTA (standard of care)

SUMMARY:
Lower extremity peripheral arterial disease is a major health problem. Currently, balloon angioplasty represents the most commonly performed treatment for patients affected by vascular claudication or critical limb ischemia. Pre-operative planning for aorto-iliac-femoral-popliteal atherosclerotic disease is a complex procedure, since an inappropriate strategy may lead to peri-operative complications. The aim of this study is to propose an innovative planning strategy for balloon angioplasty with the support of complex 3D printed models. The goal is to reduce peri-operative complications and overall costs, while improving technical success and mid-term patency of revascularizations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 89 years;
* Severe claudication or critical limb ischemia (Rutherford categories 3-5 [Cronenwett and Johnston. Rutherford's Vascular Surgery 7th edition. Saunders Elsevier 2010]) and indication already established for endovascular revascularization treatment (according to the current Italian SICVE guidelines);
* Atherosclerotic disease involving the aorto-iliac-femoro-popliteal segment;
* Signed informed consent.

Exclusion Criteria:

* Age <18 years or >89 years;
* Preoperative CTA not available for any reason (clinical contraindication, logistical impossibility);
* Patients requiring urgent intervention (lack of time for 3D model printing);
* Atherosclerotic disease limited to tibial vessels only (absent or non-significant atherosclerosis at aorto-iliac-femoro-popliteal level);
* Patient refusal to participate in the study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Confirm the effectiveness of 3D-printed models for the preoperative planning of aorto-iliac-femoral-popliteal PTA | From treatment to the end of the post-operative period (30 days)

SECONDARY OUTCOMES:
Determine the usefulness of 3D-printed models in the mid-term and during follow-up after PTA | From 1-month follow-up to 18-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria di Parma, Parma, PR, Italy

IPD SHARING:
Plan to Share IPD: No